CLINICAL TRIAL: NCT02353000
Title: Whole Brain Radiotherapy vs. Stereotactic Radiosurgery for 4 - 10 Brain Metastases:a Phase III Randomized Multicenter Trial
Brief Title: Whole Brain Radiotherapy (WBRT) Versus Stereotactic Radiosurgery (SRS) for 4 Upto 10 Brain Metastases
Acronym: WBRTvsSRS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to achieve accrural within anticipated timeframe
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-2015
Record Dates: First submitted 2015-01-16; First posted 2015-02-02 (Estimated); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Neoplasm Metastasis
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stereotactic Radiosurgery (Experimental): Stereotactic Radiosurgery for patients with 4 up to 10 brain metastases:
  Interventions: Radiation: Stereotactic Radiosurgery
- Whole Brain Radiotherapy (Other): Whole Brain Radiotherapy for patients with 4 up to 10 brain metastases:
  Interventions: Radiation: Whole Brain Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery — Stereotactic Radiosurgery for patients with 4 up to 10 brain metastases
  Arms: Stereotactic Radiosurgery
Radiation: Whole Brain Radiotherapy — Whole Brain Radiotherapy for patients with 4 up to 10 brain metastases
  Arms: Whole Brain Radiotherapy

SUMMARY:
Recently stereotactic radiosurgery (SRS) in 5 up to 10 brain metastases showed to have equal survival as in 2 up to 4 brain metastases. Whole brain radiotherapy (WBRT) is currently the gold standard for patients with more than 3 brain metastases, but has significant side effects. In this prospective randomized phase III trial WBRT is compared to SRS for patients with 4 up to 10 BM.

DETAILED DESCRIPTION:
Dutch guideline advices stereotactic radiosurgery (SRS) for patients with 1 up to 3 brain metastases (BM) and whole brain radiotherapy (WBRT) for patients with 4 or more BM. The interim analysis from the QUARTZ study showed that WBRT did not provide benefit in quality of life nor survival over best supportive care. WBRT has significant side effects, such as hair loss, fatigue, and cognitive dysfunction which may impair quality of life. A recently published study showed that SRS in patients with 5 up to 10 BM had a comparable survival to patients treated with 2 up to 4 BM. Many systemic therapies do not have a satisfactory intracranial response, because of the blood-brain barrier. The potential advantages of SRS i.e, limiting radiation doses to the uninvolved brain and a high rate of local tumour control by just a single treatment. Next logic step would be to compare WBRT with SRS alone in patients with 4-10 BM and evaluate whether SRS is superior to WBRT with regard to QOL.

ELIGIBILITY:
Inclusion Criteria:

* Minimal 4 up to a maximum of 10 BM on diagnostic MRI scan
* Max diameter of single GTV 2.5cm
* Max cumulative GTV of 30cm3
* Karnofsky performance status ≥ 70
* Any solid primary tumour. Small cell lung carcinoma, germinoma, and lymphoma are excluded
* Ability to provide written informed consent

Exclusion Criteria:

* Contra-indication for MRI
* Prior treatment for BM (i.e. surgery, SRS or WBRT)
* Concurrent use of systemic therapy
* Maximum cumulative GTV of more than 30cm3 on planning-MRI
* More than 10 BM on planning-MRI
* A brainstem metastasis with a PTV of more than 20 cm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-07; Primary Completion 2019-04 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Quality of life in patients with 4 - 10 brain metastases comparing WBRT and SRS | Change in quality of life measured from baseline to 3 months after radiotherapy
  Quality of life is measured by the EQ-5D-5L, a descriptive system of health-related quality of life states consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression)

SECONDARY OUTCOMES:
Overall survival steroid use (mg), toxicity including hair loss and fatigue. | 1 year
  Overall survival
Time that patient is functioning independently (Karnofsky ≥ 70) | Change in Karnofsky index from baseline to 3 months after radiotherapy
  Time that patient is functioning independently (Karnofsky ≥ 70)
Steroid use | Change in steroid use from baseline to 3 months after radiotherapy
  Steroid use in mg over time
Toxicity measured by hair loss and fatigue | Change in toxicity from baseline to 3 months after radiotherapy
  Toxicity measured by hair loss and fatigue using CTCAE version 4.0
Degree of independence | Change in independence from baseline to 3 months after radiotherapy
  Degree of independence of patients using the Barthel index

OTHER OUTCOMES:
Brain salvage during follow-up | 1 year
  Brain salvage during follow-up, type of salvage, and time to salvage after randomisation
Verbal learning | Change in verbal recall and verbal recognition from baseline to 3 months after radiotherapy
  Verbal recall and verbal regognition is measured using the Hopkins Verbal Learning Test - Revised
Quality of life of cancer patients | Change in Quality of life from baseline to 3 months after radiotherapy
  QoL will be measured using the EORTC QLQ-C30
Quality of life of cancer patients with brain neoplasms | Change in Quality of life from baseline to 3 months after radiotherapy
  QoL will be measured using the EORTC QLQ-BN20
Quality of life of cancer patients measuring cancer-related fatigue | Change in Quality of life from baseline to 3 months after radiotherapy
  QoL will be measured using the EORTC QLQ-FA13

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lambin, Prof. Dr., Principal Investigator — Maastro Clinic, The Netherlands
Locations (7):
- Netherlands (7):
  - VUmc, Amsterdam
  - AMC, Amsterdam
  - ZRTI, Flushing
  - Maastricht Radiation Oncology (MAASTRO clinic), Maastricht
  - Erasmus MC, Rotterdam
  - Haaglanden MC, The Hague
  - Instituut Verbeeten, Tilburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gijtenbeek JM, Ho VK, Heesters MA, Lagerwaard FJ, de Graeff A, Boogerd W. [Practice guideline 'Brain metastases' (revision)]. Ned Tijdschr Geneeskd. 2011;155(52):A4141. Dutch. PMID 22217243
- [Result] Yamamoto M, Serizawa T, Shuto T, Akabane A, Higuchi Y, Kawagishi J, Yamanaka K, Sato Y, Jokura H, Yomo S, Nagano O, Kenai H, Moriki A, Suzuki S, Kida Y, Iwai Y, Hayashi M, Onishi H, Gondo M, Sato M, Akimitsu T, Kubo K, Kikuchi Y, Shibasaki T, Goto T, Takanashi M, Mori Y, Takakura K, Saeki N, Kunieda E, Aoyama H, Momoshima S, Tsuchiya K. Stereotactic radiosurgery for patients with multiple brain metastases (JLGK0901): a multi-institutional prospective observational study. Lancet Oncol. 2014 Apr;15(4):387-95. doi: 10.1016/S1470-2045(14)70061-0. Epub 2014 Mar 10. PMID 24621620
- [Result] Zindler JD, Rodrigues G, Haasbeek CJ, De Haan PF, Meijer OW, Slotman BJ, Lagerwaard FJ. The clinical utility of prognostic scoring systems in patients with brain metastases treated with radiosurgery. Radiother Oncol. 2013 Mar;106(3):370-4. doi: 10.1016/j.radonc.2013.01.015. Epub 2013 Mar 20. PMID 23522151
- [Result] Langley RE, Stephens RJ, Nankivell M, Pugh C, Moore B, Navani N, Wilson P, Faivre-Finn C, Barton R, Parmar MK, Mulvenna PM; QUARTZ Investigators. Interim data from the Medical Research Council QUARTZ Trial: does whole brain radiotherapy affect the survival and quality of life of patients with brain metastases from non-small cell lung cancer? Clin Oncol (R Coll Radiol). 2013 Mar;25(3):e23-30. doi: 10.1016/j.clon.2012.11.002. Epub 2012 Dec 2. PMID 23211715
- [Derived] Hartgerink D, Bruynzeel A, Eekers D, Swinnen A, Hurkmans C, Wiggenraad R, Swaak-Kragten A, Dieleman E, van der Toorn PP, van Veelen L, Verhoeff JJC, Lagerwaard F, de Ruysscher D, Lambin P, Zindler J. Quality of life among patients with 4 to 10 brain metastases after treatment with whole-brain radiotherapy vs. stereotactic radiotherapy: a phase III, randomized, Dutch multicenter trial. Ann Palliat Med. 2022 Apr;11(4):1197-1209. doi: 10.21037/apm-21-1545. Epub 2021 Nov 18. PMID 34806396
- [Derived] Zindler JD, Bruynzeel AME, Eekers DBP, Hurkmans CW, Swinnen A, Lambin P. Whole brain radiotherapy versus stereotactic radiosurgery for 4-10 brain metastases: a phase III randomised multicentre trial. BMC Cancer. 2017 Jul 25;17(1):500. doi: 10.1186/s12885-017-3494-z. PMID 28743240